CLINICAL TRIAL: NCT05906732
Title: A Phase 1b/2a, 2-Part Study; Part 1: Randomized, Double-Blind, Crossover, Dose-Escalation, Placebo-Controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of SGK-1 Kinase Inhibition by LQT-1213 on Dofetilide-Induced QTc Prolongation in Healthy Adult Subjects. Part 2: Single-Blind, Multiple-Dose, Safety Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of LQT-1213 in Patients Diagnosed With Type 2 or 3 Long QT Syndrome
Brief Title: Study of LQT-1213 on QTc-induced Prolongation in Healthy Adult Subjects (Part1) and on Congenital Long QT in Patients Diagnosed With Type 2 or 3 Long QT Syndrome (Part 2).
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Advancing an alternative SGK1 inhibitor.
Sponsor: Thryv Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: LQT-1213-0061
Record Dates: First submitted 2023-06-07; First posted 2023-06-18 (Actual); Results first posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Long QT Syndrome
Keywords: LQT-1213; Congenital Long QT Syndrome; LQTS; Serum glucocorticoid regulated kinase-1; SGK-1 inhibitor; Drug induced long QT
MeSH Terms: conditions — Long QT Syndrome | interventions — dofetilide; Capsules

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1: Arm A: Dofetilide with dose-escalating LQT-1213 TID followed by Dofetilide with placebo (Experimental): Sequence A :Dofetilide 500 μg BID (Days 1-8) and LQT-1213 TID 0.25 mg/kg (Days 3 and 4), 0.50 mg/kg (Days 5 and 6), and 0.70 mg/kg on Days 7 and 8. After adequate washout, Dofetilide 500 μg BID (Days 1-8) and placebo (Days 3-8).
  Interventions: Drug: LQT-1213; Drug: Placebo; Drug: Dofetilide 250 μg Cap
- Part 1: Arm B: Dofetilide with placebo followed by Dofetilide with LQT-1213 TID (Experimental): Sequence B : Dofetilide 500 μg BID, orally (Days 1-8) and placebo TID (Days 3-8). After adequate washout, Dofetilide 500 μg BID, orally (Days 1-8) and LQT-1213 3 times a day (TID) 0.25 mg/kg (Days 3 and 4), 0.50 mg/kg (Days 5 and 6), and 0.70 mg/kg on Days 7 and 8.
  Interventions: Drug: LQT-1213; Drug: Placebo; Drug: Dofetilide 250 μg Cap
- Part 2: TID dosing of LQT-1213 16 mg (48 mg Daily) (Experimental): LQT-1213 16 mg TID (at time 0, 8 and 16 hours) on Days 2-4, with a final single morning dose on Day 4. Day 1 was placebo.
  Interventions: Drug: LQT-1213; Drug: Placebo
- Part 2: TID dosing of LQT-1213 7mg (21 mg Daily) (Experimental): LQT-1213 7 mg TID (at time 0, 8 and 16 hours) on Days 2-4, with a final single morning dose on Day 4. Day 1 was placebo.
  Interventions: Drug: LQT-1213; Drug: Placebo

INTERVENTIONS:
Drug: LQT-1213 — LQT-1213 is a serum glucocorticoid regulated kinase 1 (SGK-1) inhibitor
Drug: Placebo — Matching Placebo
Drug: Dofetilide 250 μg Cap — Dofetilide is a potent, pure inward-rectifier potassium channels (IKr) blocker
  Arms: Part 1: Arm A: Dofetilide with dose-escalating LQT-1213 TID followed by Dofetilide with placebo; Part 1: Arm B: Dofetilide with placebo followed by Dofetilide with LQT-1213 TID

SUMMARY:
Part 1: This is a Phase 1b, randomized, double-blind, crossover, dose escalation, placebo-controlled study to evaluate the effect of oral LQT-1213 on dofetilide-induced QTc prolongation in healthy adult subjects. This is a 2-treatment, 2-period crossover study with approximately up to 28 healthy subjects, with screening procedures within 28 days of enrolment.

Part 2: This is a Phase 2a, single-blind, placebo run-in, multiple-dose safety study to evaluate the safety, tolerability, and PK of LQT-1213 in patients diagnosed with LQT2 or LQT3. Up to 12 participants with LQT2 and up to 12 participants with LQT3 will be recruited.

DETAILED DESCRIPTION:
Part 1: This is a 2-treatment, 2-period crossover study. Approximately 28 healthy subjects, with the attempt to balance for sexes, will be enrolled to complete approximately up to 20 subjects in the study. In both treatment periods, all subjects will receive dofetilide on Days 1 and 2 of each period. Randomization will take place before Day 3 of Period 1. Subjects will be randomly assigned to 1 of 2 treatment sequences (AB or BA).

Part 2: Up to 12 participants with LQT2 and up to 12 participants with LQT3 will be enrolled. After initial screening, which may be conducted remotely by the CRU, individual participants with LQT2 or LQT3 will undergo a 1-day, single-blind placebo run-in period followed by 3 dosing days of LQT-1213 administered TID (the last dosing day will have a single dose). Participants will be discharged from the CRU on Day 5. Approximately 7 days after discharge from the CRU, the Follow-up Visit will be conducted remotely via telephone call.

ELIGIBILITY:
Inclusion Criteria:

Part1:

1. Male and female subjects between 18 and 60 years of age (inclusive) at Screening.
2. Not previously enrolled in a clinical study with LQT-1213.
3. Normal general health.
4. Body mass index within 18.0 to 32.0 kg/m2, inclusively at Screening.
5. Female subjects of nonchildbearing potential must be either surgically sterile (hysterectomy, bilateral tubal ligation, salpingectomy, and/or bilateral oophorectomy at least 26 weeks before Screening) or postmenopausal, defined as spontaneous amenorrhea for at least 2 years, with follicle-stimulating hormone in the postmenopausal range at Screening, based on the central laboratory's ranges.
6. Female subjects of childbearing potential (ie, ovulating, premenopausal, and not surgically sterile) must use a highly effective contraceptive regimen during their participation in the study and for 30 days after the last administration of study drug. Highly effective contraceptive methods are defined as those with <1% failure rate per year. Acceptable methods of contraception for female subjects enrolled in the study include the following:

   * Combined (estrogen- and progestogen-containing) hormonal contraception associated with inhibition of ovulation: oral, intravaginal, transdermal
   * Progestogen-only hormonal contraception associated with inhibition of ovulation: oral, injectable, implantable
   * Intrauterine device
   * Intrauterine hormone-releasing system
   * Bilateral tubal occlusion
   * Vasectomized partner
   * Heterosexual abstinence
7. Male subjects and their partners must use highly effective methods of contraception (ie, condom and spermicide) for the entire duration of the study. Male subjects must continue to use contraception and refrain from fathering a child and sperm donation for 90 days after the last administration of study drug. Acceptable methods of contraception for male subjects enrolled in the study include the following:

   * Condoms and spermicide
   * Surgical sterilization (vasectomy) of the subject at least 26 weeks before Screening
   * Heterosexual abstinence (subject must agree to use condom and spermicide if they become sexually active)
8. Understand the requirements of the study and voluntarily consent to participate in the study.

Part 2:

1. Male and female participants 18 years of age or older at Screening.
2. Body weight of at least 45 kg at Screening.
3. Female participants of nonchildbearing potential must be either surgically sterile (hysterectomy, bilateral tubal ligation, salpingectomy, and/or bilateral oophorectomy at least 26 weeks before Screening) or postmenopausal, defined as spontaneous amenorrhea for at least 2 years, with follicle-stimulating hormone in the postmenopausal range (>40 mlU/mL) at Screening, based on the central laboratory's ranges.
4. Female participants of childbearing potential (ie, ovulating, premenopausal, and not surgically sterile) must use a highly effective contraceptive regimen during their participation in the study and for 30 days after the last administration of study drug. Highly effective contraceptive methods are defined as those with <1% failure rate per year. Acceptable methods of contraception for female participants enrolled in the study include the following:

   * Combined (estrogen- and progestogen-containing) hormonal contraception associated with inhibition of ovulation: oral, intravaginal, transdermal
   * Progestogen-only hormonal contraception associated with inhibition of ovulation: oral, injectable, implantable
   * Intrauterine device
   * Intrauterine hormone-releasing system
   * Bilateral tubal occlusion
   * Vasectomized partner
   * Heterosexual abstinence
5. Male participants and their partners must use highly effective methods of contraception (ie, condom and spermicide) for the entire duration of the study. Male participants must continue to use contraception and refrain from fathering a child and sperm donation for 90 days after the last administration of study drug. Acceptable methods of contraception for male participants enrolled in the study include the following:

   * Condoms and spermicide
   * Surgical sterilization (vasectomy) of the participant at least 26 weeks before Screening
   * Heterosexual abstinence (participant must agree to use condom and spermicide if they become sexually active)
6. LQT2 or LQT3 mutation:

   * LQTS 2: Participants with potassium voltage-gated channel subfamily H member 2 (KCNH2) mutations that are dominant negative and considered to be pathologic or likely pathologic by the screening laboratory can be included after approval from the sponsor. Participants with haploinsufficiency will not be eligible for this study.
   * LQTS 3: Participants with a sodium voltage-gated channel alpha subunit 5 (SCN5A) gene chromosome 3 mutations that are mutations and considered to be pathologic or likely pathologic by the screening laboratory can be included after approval from the sponsor. Participants with mutations not associated with Brugada syndrome or overlap syndromes or where mutations affect the window current or the persistent 'late' Na current to exert a primary or major role in the phenotype, will be eligible for this study.
7. QTcF interval ≥480 and ≤560 ms determined at Screening and on Day -1 triplicate ECGs as assessed by a physician trained in complex ECG interpretation.
8. The first 2 participants with LQT2 require having an ICD before further participants with LQT2 are enrolled and the first 2 participants with LQT3 require having an ICD before further participants with LQT3 are enrolled. This stipulation may be altered based on agreement between the principal investigator and Sponsor based on emerging data. The ICD implantation must have been at least 2 months before Screening.

   Note: Subsequent participants may or may not have had an ICD. The results of the ICD interrogation within the last 6 months should be available for review unless waived by the investigator and sponsor.
9. Understand the requirements of the study and voluntarily consent to participate in the study.

Exclusion Criteria:

Part 1:

1. On Day 1 at 3 hours postdose in Period 1 only, of the first cycle of dofetilide, the QTcF on the triplicate ECGs will be manually confirmed by cardiologist experienced in ECG interval measurements. The ECG measurements at baseline and at the 3-hour time points will be performed by the same technician and cardiologist. If the mean QTcF increase from baseline is <25 ms on triplicate safety ECGs compared to the mean from baseline (all ECG QTcF measurements averaged), the subject will be disqualified from further study participation.
2. Clinically significant gastrointestinal, renal, hepatic, neurologic, hematologic, endocrine, oncologic, pulmonary, immunologic, psychiatric, or cardiovascular disease or any other condition, which, in the opinion of the investigator, would jeopardize the safety of the subject or impact the validity of the study results. No history of myocardial infarction or angina or ischemic heart disease, nonsustained or sustained ventricular tachycardia, atrial fibrillation, stroke, transient ischemic attack, syncope, congestive heart failure, family history of LQTS, Torsades de Pointes, or sudden cardiac death.
3. Female subjects must not be pregnant, lactating, or breastfeeding, and must not be planning to become pregnant.
4. Female subjects of childbearing potential must have a negative result for the serum pregnancy test at Screening and Check-in.
5. Clinically significant abnormal findings on the physical examination or medical history during Screening as deemed by the investigator.
6. Participated in a previous clinical study in the previous 3 months before dosing.
7. Donation of blood volume greater than 300 mL within 30 days before Screening and agree to avoid donation from Screening and throughout the study.
8. At Screening and on Day -2, if the 12-lead ECG demonstrates any of the following: PR >240 ms; QRS >110 ms, or QTcF <400 ms and >440 ms; second- or third-degree atrioventricular block; bundle branch block, significant ST-T wave abnormalities or flat T waves that could interfere with QT analysis. If HR <50 or >85 bpm, then 2 more ECGs will be recorded, and the mean values will be used.
9. Known sensitivity to kinase inhibitors.
10. Abnormal renal function with an estimated glomerular filtration rate (eGFR) of <70 mL/min/1.73 m2, with eGFR calculated by the Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] formula at Screening. One retest of the exclusionary eGFR value is allowed at the discretion of the investigator.
11. Subject has abnormal liver function tests (transaminases or total bilirubin) greater than 2.5 × the upper limit of normal at Screening or baseline. One retest of exclusionary abnormal liver function tests is allowed at the discretion of the investigator.
12. Subject has a positive serology test for HIV antibodies, hepatitis B surface antigen, or hepatitis C virus antibody at Screening.
13. Subject has a hemoglobin <11.0 g/dL, potassium <3.8 mg/dL, magnesium <1.9 mg/dL, or calcium <8.5 mg/dL at Screening or baseline. One retest of exclusionary hemoglobin, potassium, magnesium, and calcium is allowed at the discretion of the investigator. Electrolyte supplementation is allowed at any time as long as it is >4 hours before dosing.
14. Subject has a history of hypersensitivity to drugs with a clinically significant reaction or any clinically significant hypersensitivities.
15. Subject has an allergy to band aids, adhesive dressing, or medical tape.
16. Subject has a history within the past 2 months of strenuous exercise (eg, marathon running) and is unwilling to refrain from strenuous exercise from 7 days before Check-in and until the end of the study. Subject has abnormal creatine phosphokinase test greater than 3 × the upper limit of normal at Screening and baseline. One retest of exclusionary abnormal creatine phosphokinase tests is allowed at the discretion of the investigator.
17. Subject is unable to refrain from or anticipates the use of any drug, including prescription and nonprescription medications (with the exception of hormonal contraception), herbal preparations, or vitamin supplements beginning 14 days before the first dose and until the end of the study. After dosing, acetaminophen (up to 2 g per 24 hours) may be administered at the discretion of the investigator or designee.

    1. Hepatic or renal clearance altering agents within 30 days before the first dose and until the end of the study.
    2. Avoid vaccinations from Screening until the end of the study.
    3. Has consumed cruciferous vegetables (eg, kale, broccoli, watercress, collard greens, kohlrabi, Brussels sprouts, and mustard greens) or charbroiled meats within 7 days before Check-in through the Follow-up Visit.
    4. Use of any drugs known to be significant strong inducers of cytochrome P450 (CYP) 3A enzymes, including St. John's Wort, for 28 days before Day -1 or 5 half-lives (whichever is longer) and through the Follow-up Visit.
    5. Has consumed Seville oranges, grapefruit and/or grapefruit juice within 14 days before Check-in and is unwilling to abstain from consuming these items until the end of the study.
18. Subject is considering or scheduled to undergo any surgical procedure during the study.
19. Subject has experienced an acute illness that has resolved in less than 14 days before the first study drug dose or has had a major illness or hospitalization within 1 month before the first study drug dose.
20. Subject is unwilling to abstain from ingestion of caffeine- or xanthine-containing products (eg, tea, coffee, chocolate, cola, etc.) beginning 96 hours before Check-in until the final PK sample of the study has been collected.
21. Subject is unwilling to abstain from alcohol beginning 48 hours before Check-in and until the final PK sample of the study has been collected.
22. Subject has a history of high alcohol consumption within 9 months before Screening, defined as an average weekly intake of >14 units for males or >10 units for females.

    One unit is equivalent to 8 g of alcohol: a half-pint (~240 mL) of beer, 1 glass (125 mL) of wine, or 1 measure (25 mL) of spirits.
23. Subject has a history of drug abuse in the 3 years before Screening or positive screen for drugs of abuse or alcohol at Screening or baseline. Subjects may undergo a repeat urine drug screen at the discretion of the investigator.
24. Subject uses or has used tobacco-or nicotine-containing products (eg, cigarettes, cigars, chewing tobacco, snuff, etc.) within 6 months before Screening and is unwilling to abstain from tobacco-containing products until the end of the study, based on subject self-reporting.
25. Subject, who, for any reason, is deemed by the investigator to be inappropriate for this study or has any condition which would confound or interfere with the evaluation of the safety, tolerability, or PK of the investigational drug or prevent compliance with the study protocol.

Part 2:

1. Clinically significant gastrointestinal, renal, hepatic, neurologic, hematologic, endocrine, oncologic, pulmonary, immunologic, psychiatric, or significant structural cardiovascular disease or any other condition beyond LQT2 or LQT3, which, in the opinion of the investigator or sponsor, would jeopardize the safety of the participant or impact the validity of the study results. History of myocardial infarction or ongoing angina or active ischemic heart disease, atrial fibrillation, stroke, or transient ischemic attack within the past 12 months, greater than New York Heart Association Class II congestive heart failure, bundle branch block, hemodynamically significant ventricular tachycardia not due to Torsades de Pointes, or Brugada syndrome.
2. Participant has a history of an aborted cardiac arrest, ICD implantation, syncopal episode due to a ventricular arrhythmia or where confidence in the etiology cannot be established, or appropriate ICD therapy for ventricular tachycardia/ventricular fibrillation within 2 months before Screening. Participants with LQT2 or LQT3 can be enrolled after the 2-month time period has lapsed.
3. Female participants must not be pregnant, lactating, or breastfeeding, and must not be planning to become pregnant.
4. Female participants of childbearing potential must have a negative result for the serum pregnancy test at Screening and Check-in.
5. Clinically significant abnormal findings on the physical examination at Check-in or medical history during Screening as deemed by the principal investigator.
6. Currently participating in another interventional clinical study.
7. Donation of blood volume greater than 300 mL within 30 days before dosing and unwilling to avoid donation from Screening and throughout the study.
8. Screening diastolic blood pressure <45 or >95 mm Hg, systolic blood pressure <90 or >150 mm Hg, or with sponsor and investigator approval.
9. At Screening and on Day -1, if the triplicate 12-lead ECG demonstrates any of the following: mean PR >250ms; QRS >110 ms, or QTcF >560 ms and <480 ms; bundle branch block or significant ST-T wave abnormalities or flat T waves that could interfere with QT analysis. Heart rate <45 bpm, unless receiving a beta-blocker in which case <40 bpm, or HR >95 bpm. If any of these exclusionary criteria are met, then a second set of triplicate ECGs may be acquired, and the mean values may be used. For participants on beta blockade, the PR interval may be higher than 250 ms with sponsor and investigator approval.
10. Atrial pacing rate set to ≥80 bpm in those with atrial pacing.
11. Participant has a pacemaker or ICD that is actively used for ventricular pacing.
12. Known sensitivity to kinase inhibitors or clinically significant drug allergies to any of the components of LQT-1213.
13. Abnormal renal function with an eGFR of <60 mL/min/1.73 m2, with eGFR calculated by the CKD-EPI formula at Screening. One retest of the exclusionary eGFR value is allowed at Screening and Check-in at the discretion of the investigator.
14. Participant has abnormal liver function tests (transaminases greater than 2 × the upper limit of normal [ULN] or total bilirubin > 1.5 × ULN. If the participant has documented Gilbert's Syndrome, participation is at the combined principal investigator and Sponsor's discretion after review of historical liver and bilirubin tests.
15. Participant has a positive serology test for HIV antibodies, hepatitis B surface antigen, or hepatitis C virus antibody at Screening.
16. Participant has a hemoglobin <11.0 g/dL, potassium <3.8 mg/dL, magnesium <1.8 mg/dL, or calcium <8.5 mg/dL at Screening or baseline. One retest of exclusionary hemoglobin, potassium, magnesium, and calcium is allowed at the discretion of the investigator.
17. Participant has a history of hypersensitivity to drugs with a clinically significant reaction or any clinically significant hypersensitivities.
18. Participant has a clinically significant allergy to band aids, adhesive dressing, ECG electrodes, or medical tape.
19. Participant has abnormal creatine phosphokinase test greater than 3 × the ULN at Screening or baseline. One retest of exclusionary abnormal creatine phosphokinase tests is allowed at the discretion of the investigator.
20. Participant is currently taking, within the last 7 days before Spaulding admission or 5 half-lives (whichever is longer), or anticipates the use of any antiarrhythmic medications (including mexilitene except beta-blockers which are allowed,) or drugs known to affect the QT interval (including ranolazine; refer to drug lists for "Drugs with known, possible, or conditional risk of TdP" that are known to prolong the QT interval at https://crediblemeds.org), unless approved by the sponsor and principal investigator.
21. Participant is not permitted to use/consume the following:

    1. Any drugs known to be significant strong inducers of CYP 3A enzymes, including St. John's Wort, for 28 days before Day -1 or 5 half-lives (whichever is longer) and through the Follow-up Visit.
    2. Seville oranges, grapefruit and/or grapefruit juice within 7 days before Check-in and is unwilling to abstain from consuming these items until the end of the study.
22. Participant is considering or scheduled to undergo any surgical procedure during the study.
23. Participant has experienced an acute illness that has resolved in less than 14 days before the first study drug dose or has had a major illness or hospitalization within 1 month before the first study drug dose.
24. Participant is unwilling to abstain from ingestion of caffeine- or xanthine-containing products (eg, tea, coffee, chocolate, cola, etc.) beginning 96 hours before Check-in until the final PK sample of the study has been collected.
25. Participant is unwilling to abstain from alcohol beginning 48 hours before Check-in and until the final PK sample of the study has been collected.
26. Participant has a history of high alcohol consumption or substance abuse that would pose a risk for the participant's safety and compliance with the study protocol. Participant must not have positive screen for drugs of abuse at Screening or baseline and alcohol at baseline, except with sponsor permission. Participants may undergo a repeat urine drug screen at the discretion of the investigator.
27. Participant, who, for any reason, is deemed by the investigator to be inappropriate for this study or has any condition which would confound or interfere with the evaluation of the safety, tolerability, or PK of the investigational drug or prevent compliance with the study protocol.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2023-03-12 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Matousek, DO, Principal Investigator — Spaulding Clinical Research LLC
Locations (1):
- Spaulding Clinical Research, LLC, West Bend, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Part 1: Arm A: Dofetilide With Dose-escalating LQT-1213 TID Followed by Dofetilide With Placebo: Dofetilide 500 μg BID (Days 1-8) and LQT-1213 TID 0.25 mg/kg (Days 3 and 4), 0.50 mg/kg (Days 5 and 6), and 0.70 mg/kg on Days 7 and 8. After adequate washout, Dofetilide 500 μg BID (Days 1-8) and placebo (Days 3-8).
  LQT-1213: LQT-1213 is a serum glucocorticoid regulated kinase 1 (SGK-1) inhibitor
  Placebo: Matching Placebo
  Dofetilide 250 μg Cap: Dofetilide is a potent, pure inward-rectifier potassium channels (IKr) blocker
- Part 1: Arm B: Dofetilide With Placebo Followed by Dofetilide With LQT-1213 TID: Dofetilide 500 μg BID, orally (Days 1-8) and placebo matched to LQT-1213 TID (Days 3-8). After adequate washout, Dofetilide 500 μg BID, orally (Days 1-8) and LQT-1213 3 times a day (TID) 0.25 mg/kg (Days 3 and 4), 0.50 mg/kg (Days 5 and 6), and 0.70 mg/kg on Days 7 and 8.
  LQT-1213: LQT-1213 is a serum glucocorticoid regulated kinase 1 (SGK-1) inhibitor
  Placebo: Matching Placebo
  Dofetilide 250 μg Cap: Dofetilide is a potent, pure inward-rectifier potassium channels (IKr) blocker
- Part 2: TID Dosing of LQT-1213 7 mg (21 mg Daily): LQT-1213 7 mg TID (at time 0, 8 and 16 hours) on Days 2-4, with a final single morning dose on Day 4. Day 1 was placebo.
  LQT-1213: LQT-1213 is a serum glucocorticoid regulated kinase 1 (SGK-1) inhibitor
  Placebo: Matching Placebo
Period: Overall Study
Arm/Group | Part 1: Arm A: Dofetilide With Dose-escalating LQT-1213 TID Followed by Dofetilide With Placebo | Part 1: Arm B: Dofetilide With Placebo Followed by Dofetilide With LQT-1213 TID | Part 2: TID Dosing of LQT-1213 16 mg (48 mg Daily) | Part 2: TID Dosing of LQT-1213 7 mg (21 mg Daily)
Started | 15 | 15 | 6 | 6
Completed | 12 | 11 | 6 | 6
Not Completed | 3 | 4 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — Physician Decision | 2 | 4 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part 2: TID Dosing of LQT-1213 16 mg: LQT-1213 16 mg TID (at time 0, 8 and 16 hours) on Days 2-4, with a final single morning dose on Day 4. Day 1 was placebo.
  LQT-1213: LQT-1213 is a serum glucocorticoid regulated kinase 1 (SGK-1) inhibitor
  Placebo: Matching Placebo
- Part 2: TID Dosing of LQT-1213 7mg: LQT-1213 7 mg TID (at time 0, 8 and 16 hours) on Days 2-4, with a final single morning dose on Day 4. Day 1 was placebo.
  LQT-1213: LQT-1213 is a serum glucocorticoid regulated kinase 1 (SGK-1) inhibitor
  Placebo: Matching Placebo
- Total: Total of all reporting groups
Arm/Group | Part 1: Arm A: Dofetilide With Dose-escalating LQT-1213 TID Followed by Dofetilide With Placebo | Part 1: Arm B: Dofetilide With Placebo Followed by Dofetilide With LQT-1213 TID | Part 2: TID Dosing of LQT-1213 16 mg | Part 2: TID Dosing of LQT-1213 7mg | Total
Number analyzed (Participants) | 15 | 15 | 6 | 6 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.3 (12.4) | 42.2 (9.13) | 42.0 (13.71) | 40.3 (8.33) | 42 (10.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 4 | 5 | 18
  Male | 10 | 11 | 2 | 1 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 2 | 0 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 8 | 6 | 0 | 0 | 14
  White | 6 | 7 | 6 | 6 | 25
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
body mass index [Mean (Standard Deviation); unit: kg/m2] | 27.35 (3.365) | 26.99 (2.942) | 30.82 (6.971) | 33.33 (7.560) | 28.57 (4.33)

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Pharmacodynamics: By-time Point Analysis for QTc on LQT-1213 Versus Placebo
Description: The primary outcome is time-based comparison in the change from baseline (baseline defined as Day 1 of Period 1 and Day 1 of Period 2 mean predose QTc) ΔΔQTc by Fridericia's formula (QTcF) during peak dofetilide exposure between dofetilide and placebo treatment, and the dofetilide and LQT-1213 treatment.
Time Frame: 2.0 hours after administration of study treatment on Day 4.
Population: All subjects who received at least 1 dose of any study treatment (dofetilide, LQT-1213, or placebo) and had measurements at baseline as well as on-treatment with at least 1 post-baseline time point with a ΔQTc value.
Measure: Mean (Standard Error); unit: msec
Groups:
- Dofetilide + LQT-1213 0.25 mg/kg (Day 4): Dofetilide 500 μg twice a day (BID) orally (Days 1-8) and LQT-1213 three times a day (TID) 0.25 mg/kg (Days 3 and 4), mid dose (Days 5 and 6) 0.50 mg/kg and high dose (Days 7 and 8) 0.70 mg/kg.
- Dofetilide + Placebo (Day 4): Dofetilide 500 μg twice a day (BID) orally (Days 1-8) + placebo tid (Days3-8)
Arm/Group | Dofetilide + LQT-1213 0.25 mg/kg (Day 4) | Dofetilide + Placebo (Day 4)
Number analyzed (Participants) | 28 | 29
msec | 40.8 (11.08) | 50.3 (14.77)
Statistical Analysis 1: Comparison: Dofetilide + LQT-1213 0.25 mg/kg (Day 4) vs Dofetilide + Placebo (Day 4); Test type: Superiority; p = 0.0030, Mixed Models Analysis; LS Mean = -9.6

2. Primary Outcome: Part 1: Pharmacodynamics: By-time Point Analysis for QTc on LQT-1213 Versus Placebo
Description: as for outcome 1
Time Frame: 2.5 hours after administration of study treatment on Day 4
Population: as for outcome 1
Measure: Mean (Standard Error); unit: msec
Groups:
- Dofetilide + Placebo (Day 4): Dofetilide 500 μg twice a day (BID) orally (Days 1-8) and Placebo three times a day (TID) (Days 3-8)
Arm/Group | Dofetilide + LQT-1213 0.25 mg/kg (Day 4) | Dofetilide + Placebo (Day 4)
Number analyzed (Participants) | 27 | 28
msec | 43.3 (11.76) | 48.0 (11.42)
Statistical Analysis 1: Comparison: Dofetilide + LQT-1213 0.25 mg/kg (Day 4) vs Dofetilide + Placebo (Day 4); Test type: Superiority; p = 0.0266, Mixed Models Analysis; LS Mean = -6.5

3. Primary Outcome: Part 1: Pharmacodynamics: By-time Point Analysis for QTc on LQT-1213 Versus Placebo
Description: as for outcome 1
Time Frame: 3.0 hours after administration of study treatment on Day 4
Population: as for outcome 1
Measure: Mean (Standard Error); unit: msec
Groups:
- Dofetilide + Placebo (Day 4): Dofetilide 500 μg twice a day (BID) orally (Days 1-8) and Placebo tid (Days 3-8)
Arm/Group | Dofetilide + LQT-1213 0.25 mg/kg (Day 4) | Dofetilide + Placebo (Day 4)
Number analyzed (Participants) | 28 | 29
msec | 40.9 (11.05) | 48.6 (12.93)
Statistical Analysis 1: Comparison: Dofetilide + LQT-1213 0.25 mg/kg (Day 4) vs Dofetilide + Placebo (Day 4); Test type: Superiority; p = 0.0067, Mixed Models Analysis; LS Mean = -7.8

4. Primary Outcome: Part 1: Pharmacodynamics: By-time Point Analysis for QTc on LQT-1213 Versus Placebo
Description: as for outcome 1
Time Frame: 3.5 hours after administration of study treatment on Day 4
Population: as for outcome 1
Measure: Mean (Standard Error); unit: msec
Arm/Group | Dofetilide + LQT-1213 0.25 mg/kg (Day 4) | Dofetilide + Placebo (Day 4)
Number analyzed (Participants) | 28 | 28
msec | 43.4 (13.01) | 46.4 (11.33)
Statistical Analysis 1: Comparison: Dofetilide + LQT-1213 0.25 mg/kg (Day 4) vs Dofetilide + Placebo (Day 4); Test type: Superiority; p = 0.1106, Mixed Models Analysis; LS Mean = -3.9

5. Primary Outcome: Part 1: Pharmacodynamics: By-time Point Analysis for QTc on LQT-1213 Versus Placebo
Description: as for outcome 1
Time Frame: 4.0 hours after administration of study treatment on Day 4
Population: as for outcome 1
Measure: Mean (Standard Error); unit: msec
Arm/Group | Dofetilide + LQT-1213 0.25 mg/kg (Day 4) | Dofetilide + Placebo (Day 4)
Number analyzed (Participants) | 28 | 29
msec | 39.2 (10.85) | 43.3 (13.83)
Statistical Analysis 1: Comparison: Dofetilide + LQT-1213 0.25 mg/kg (Day 4) vs Dofetilide + Placebo (Day 4); Test type: Superiority; p = 0.0908, Mixed Models Analysis; LS Mean = -4.2

6. Primary Outcome: Part 1: Pharmacodynamics: By-time Point Analysis for QTc on LQT-1213 Versus Placebo
Description: as for outcome 1
Time Frame: 2.0 hours after administration of study treatment on Day 6
Population: as for outcome 1
Measure: Mean (Standard Error); unit: msec
Groups:
- Dofetilide + LQT-1213 0.50 mg/kg (Day 6): Dofetilide 500 μg twice a day (BID) orally (Days 1-8) and LQT-1213 three times a day (TID) 0.25 mg/kg (Days 3 and 4), mid dose (Days 5 and 6) 0.50 mg/kg and high dose (Days 7 and 8) 0.70 mg/kg.
- Dofetilide + Placebo (Day 6): Dofetilide 500 μg twice a day (BID) orally (Days 1-8) and Placebo TID (Days 3-8).
Arm/Group | Dofetilide + LQT-1213 0.50 mg/kg (Day 6) | Dofetilide + Placebo (Day 6)
Number analyzed (Participants) | 23 | 25
msec | 42.4 (15.89) | 43.9 (16.41)
Statistical Analysis 1: Comparison: Dofetilide + LQT-1213 0.50 mg/kg (Day 6) vs Dofetilide + Placebo (Day 6); Test type: Superiority; p = 0.4038, Mixed Models Analysis; LS Mean = -1.2

7. Primary Outcome: Part 1: Pharmacodynamics: By-time Point Analysis for QTc on LQT-1213 Versus Placebo
Description: as for outcome 1
Time Frame: 2.5 hours after administration of study treatment on Day 6
Population: as for outcome 1
Measure: Mean (Standard Error); unit: msec
Arm/Group | Dofetilide + LQT-1213 0.50 mg/kg (Day 6) | Dofetilide + Placebo (Day 6)
Number analyzed (Participants) | 23 | 26
msec | 43.7 (14.74) | 42.5 (16.93)
Statistical Analysis 1: Comparison: Dofetilide + LQT-1213 0.50 mg/kg (Day 6) vs Dofetilide + Placebo (Day 6); Test type: Superiority; p = 0.6255, Mixed Models Analysis; LS Mean = 1.5

8. Primary Outcome: Part 1: Pharmacodynamics: By-time Point Analysis for QTc on LQT-1213 Versus Placebo
Description: as for outcome 1
Time Frame: 3.0 hours after administration of study treatment on Day 6
Population: as for outcome 1
Measure: Mean (Standard Error); unit: msec
Groups:
- Dofetilide + Placebo (Day6): Dofetilide 500 μg twice a day (BID) orally (Days 1-8) and Placebo (Days 3-6)
Arm/Group | Dofetilide + LQT-1213 0.50 mg/kg (Day 6) | Dofetilide + Placebo (Day6)
Number analyzed (Participants) | 23 | 24
msec | 42.3 (12.57) | 40.4 (16.70)
Statistical Analysis 1: Comparison: Dofetilide + LQT-1213 0.50 mg/kg (Day 6) vs Dofetilide + Placebo (Day6); Test type: Superiority; p = 0.5140, Mixed Models Analysis; LS Mean = 0.2

9. Primary Outcome: Part 1: Pharmacodynamics: By-time Point Analysis for QTc on LQT-1213 Versus Placebo
Description: as for outcome 1
Time Frame: 3.5 hours after administration of study treatment on Day 6
Population: as for outcome 1
Measure: Mean (Standard Error); unit: msec
Groups:
- LQT-1213 0.50 mg/kg (Day 6): Dofetilide 500 μg twice a day (BID) orally (Days 1-8) and LQT-1213 three times a day (TID) 0.25 mg/kg (Days 3 and 4), mid dose (Days 5 and 6) 0.50 mg/kg and high dose (Days 7 and 8) 0.70 mg/kg.
- Dofetilide + Placebo (Day 6): Dofetilide 500 μg twice a day (BID) orally (Days 1-8) and placebo (Days 3-8)
Arm/Group | LQT-1213 0.50 mg/kg (Day 6) | Dofetilide + Placebo (Day 6)
Number analyzed (Participants) | 23 | 24
msec | 42.0 (13.40) | 40.7 (15.45)
Statistical Analysis 1: Comparison: LQT-1213 0.50 mg/kg (Day 6) vs Dofetilide + Placebo (Day 6); Test type: Superiority; p = 0.5675, Mixed Models Analysis; LS Mean = 0.8

10. Primary Outcome: Part 1: Pharmacodynamics: By-time Point Analysis for QTc on LQT-1213 Versus Placebo
Description: as for outcome 1
Time Frame: 4.0 hours after administration of study treatment on Day 6
Population: as for outcome 1
Measure: Mean (Standard Error); unit: msec
Arm/Group | Dofetilide + LQT-1213 0.50 mg/kg (Day 6) | Dofetilide + Placebo (Day 6)
Number analyzed (Participants) | 24 | 27
msec | 38.5 (14.64) | 35.3 (17.14)
Statistical Analysis 1: Comparison: Dofetilide + LQT-1213 0.50 mg/kg (Day 6) vs Dofetilide + Placebo (Day 6); Test type: Superiority; p = 0.7640, Mixed Models Analysis; LS Mean = 3.4

11. Primary Outcome: Part 1: Pharmacodynamics: By-time Point Analysis for QTc on LQT-1213 Versus Placebo
Description: as for outcome 1
Time Frame: 2.0 hours after administration of study treatment on Day 8
Population: as for outcome 1
Measure: Mean (Standard Error); unit: msec
Groups:
- Dofetilide + LQT-1213 0.70 mg/kg (Day 8): Dofetilide 500 μg twice a day (BID) orally (Days 1-8) and LQT-1213 three times a day (TID) 0.25 mg/kg (Days 3 and 4), mid dose (Days 5 and 6) 0.50 mg/kg and high dose (Days 7 and 8) 0.70 mg/kg.
- Dofetilide + Placebo (Day 8): Dofetilide 500 μg twice a day (BID) orally (Days 1-8) and placebo (Days 3-8)
Arm/Group | Dofetilide + LQT-1213 0.70 mg/kg (Day 8) | Dofetilide + Placebo (Day 8)
Number analyzed (Participants) | 23 | 27
msec | 45.0 (14.31) | 48.9 (13.94)
Statistical Analysis 1: Comparison: Dofetilide + LQT-1213 0.70 mg/kg (Day 8) vs Dofetilide + Placebo (Day 8); Test type: Superiority; p = .2437, Mixed Models Analysis; LS Mean = -2.8

12. Primary Outcome: Part 1: Pharmacodynamics: By-time Point Analysis for QTc on LQT-1213 Versus Placebo
Description: as for outcome 1
Time Frame: 2.5 hours after administration of study treatment on Day 8
Population: as for outcome 1
Measure: Mean (Standard Error); unit: msec
Groups:
- LQT-1213 0.70 mg/kg (Day 8): Dofetilide 500 μg twice a day (BID) orally (Days 1-8) and LQT-1213 three times a day (TID) 0.25 mg/kg (Days 3 and 4), mid dose (Days 5 and 6) 0.50 mg/kg and high dose (Days 7 and 8) 0.70 mg/kg.
- Dofetilide + Placebo (Day 8): Dofetilide 500 μg twice a day (BID) orally (Days 1-8) and Placebo TID (Days 3-8)
Arm/Group | LQT-1213 0.70 mg/kg (Day 8) | Dofetilide + Placebo (Day 8)
Number analyzed (Participants) | 24 | 25
msec | 46.6 (14.23) | 46.8 (11.45)
Statistical Analysis 1: Comparison: LQT-1213 0.70 mg/kg (Day 8) vs Dofetilide + Placebo (Day 8); Test type: Superiority; p = 0.4229, Mixed Models Analysis; LS Mean = -0.8

13. Primary Outcome: Part 1: Pharmacodynamics: By-time Point Analysis for QTc on LQT-1213 Versus Placebo
Description: as for outcome 1
Time Frame: 3.0 hours after administration of study treatment on Day 8
Population: as for outcome 1
Measure: Mean (Standard Error); unit: msec
Arm/Group | Dofetilide + LQT-1213 0.70 mg/kg (Day 8) | Dofetilide + Placebo (Day 8)
Number analyzed (Participants) | 24 | 25
msec | 46.4 (15.18) | 48.0 (13.24)
Statistical Analysis 1: Comparison: Dofetilide + LQT-1213 0.70 mg/kg (Day 8) vs Dofetilide + Placebo (Day 8); Test type: Superiority; p = 0.4887, Mixed Models Analysis; LS Mean = -0.1

14. Primary Outcome: Part 1: Pharmacodynamics: By-time Point Analysis for QTc on LQT-1213 Versus Placebo
Description: as for outcome 1
Time Frame: 3.5 hours after administration of study treatment on Day 8
Population: as for outcome 1
Measure: Mean (Standard Error); unit: msec
Arm/Group | Dofetilide + LQT-1213 0.70 mg/kg (Day 8) | Dofetilide + Placebo (Day 8)
Number analyzed (Participants) | 24 | 26
msec | 44.4 (13.84) | 48.3 (12.34)
Statistical Analysis 1: Comparison: Dofetilide + LQT-1213 0.70 mg/kg (Day 8) vs Dofetilide + Placebo (Day 8); Test type: Superiority; p = 0.2042, Mixed Models Analysis; LS Mean = -3.1

15. Primary Outcome: Part 1: Pharmacodynamics: By-time Point Analysis for QTc on LQT-1213 Versus Placebo
Description: as for outcome 1
Time Frame: 4.0 hours after administration of study treatment on Day 8
Population: as for outcome 1
Measure: Mean (Standard Error); unit: msec
Arm/Group | Dofetilide + LQT-1213 0.70 mg/kg (Day 8) | Dofetilide + Placebo (Day 8)
Number analyzed (Participants) | 23 | 25
msec | 41.4 (12.25) | 45.7 (11.75)
Statistical Analysis 1: Comparison: Dofetilide + LQT-1213 0.70 mg/kg (Day 8) vs Dofetilide + Placebo (Day 8); Test type: Superiority; p = 0.2644, Mixed Models Analysis; Mean Difference (Net) = -2.2

16. Primary Outcome: Part 2: Safety and Tolerability of Oral LQT-1213 in Participants With LQT-2 or LQT-3
Description: The primary outcome is to measure the incidence of treatment emergent adverse events (TEAEs).
Time Frame: up to day 12
Population: all participants with LQT2, or LQT3 who received at least 1 dose of study drug (placebo or LQT-1213) and provide at least 1 postdose safety assessment.
Measure: Number; unit: TEAE
Groups:
- LQT-1213 16 mg TID (48 mg Daily): LQT-1213 16 mg TID (at time 0, 8 and 16 hours) on Days 2-4, with a final single morning dose on Day 4.
- LQT-1213 7mg Tid (21 mg Daily): LQT-1213 7 mg TID (at time 0, 8 and 16 hours) on Days 2-4, with a final single morning dose on Day 4.
- Placebo in LQT-1213 16 mg TID (48 mg): Placebo in LQT-1213 16 mg TID (48 mg) Day 1 Placebo
- Placebo in LQT-1213 7 mg TID (21 mg): Placebo in LQT-1213 7 mg TID (21 mg) - Day 1 Placebo
Arm/Group | LQT-1213 16 mg TID (48 mg Daily) | LQT-1213 7mg Tid (21 mg Daily) | Placebo in LQT-1213 16 mg TID (48 mg) | Placebo in LQT-1213 7 mg TID (21 mg)
Number analyzed (Participants) | 6 | 6 | 6 | 6
TEAE | 4 | 3 | 1 | 2

17. Secondary Outcome: Part 1: Pharmacokinetic LQT-1213 AUC0-t
Description: Area under the concentration-time curve (AUC) from time 0 to the time of the last measurable concentration
Time Frame: 0 to 24 hours post-dose on Day 8
Population: The overall number of participants analyzed for PK parameters includes all individuals who had available the PK parameter, regardless of whether this data was collected in Period 1 or Period 2 of the two sequences described in the participant Flow.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/ml
Groups:
- LQT-1213 TID 0.70 mg/kg: Dofetilide 500 μg BID, orally (Days 1-8) and LQT-1213 TID 0.25 mg/kg (Days 3 and 4), 0.50 mg/kg (Days 5 and 6), and 0.70 mg/kg on (Days 7 and 8).
Arm/Group | LQT-1213 TID 0.70 mg/kg
Number analyzed (Participants) | 25
h*ng/ml | 13221.182 (47.6)

18. Secondary Outcome: Part 1: Pharmacokinetic Dofetilide AUC0-t
Description: Area under the concentration-time curve (AUC) from time 0 to the time of the last measurable concentration
Time Frame: 0 to 24 hours post-dose on Day 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/ml
Groups:
- Dofetilide 500 μg + Placebo Day 8: Dofetilide 500 μg BID, orally (Days 1-8) combined to placebo. Single dose was given on the morning of Day 8.
- Dofetilide 500 μg + LQT-1213: Dofetilide 500 µg twice daily (BID) orally on Days 1-8 and LQT-1213 3 times a day (TID) (0, 7.75, and 17 hours) orally on Days 3-8 as low dose (0.25 mg/kg) on Day 3 through the second dose on Day 4, mid dose (0.50 mg/kg) for last dose on Day 4 through the second dose on Day 6, and high dose (0.70 mg/kg) for last dose on Day 6 through the dose on Day 8.
Arm/Group | Dofetilide 500 μg + Placebo Day 8 | Dofetilide 500 μg + LQT-1213
Number analyzed (Participants) | 25 | 25
h*ng/ml | 50.160 (18.6) | 51.863 (17.1)

19. Secondary Outcome: Part 1: Pharmacokinetic LQT-1213 AUCtau
Description: AUCtau = Area under the curve from time 0 to 8.0 hours
Time Frame: Day 4,6, 8
Population: pk population= at least 1 evaluable PK concentration for dofetilide or LQT-1213
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/ml
Groups:
- LQT-1213 0.25 mg/kg (Day 4) TID; LQT-1213 0.50 mg/kg (Day 6) TID; LQT-1213 0.70 mg/kg (Day 8) TID: Dofetilide 500 μg twice a day (BID) orally (Days 1-8) and LQT-1213 three times a day (TID) 0.25 mg/kg (Days 3 and 4), mid dose (Days 5 and 6) 0.50 mg/kg and high dose (Days 7 and 8) 0.70 mg/kg.
Arm/Group | LQT-1213 0.25 mg/kg (Day 4) TID | LQT-1213 0.50 mg/kg (Day 6) TID | LQT-1213 0.70 mg/kg (Day 8) TID
Number analyzed (Participants) | 29 | 25 | 25
h*ng/ml | 2735.793 (47.9) | 5433.729 (49.6) | 8763.318 (48.0)

20. Secondary Outcome: Part 1: Pharmacokinetic Dofetilide AUCtau
Description: AUCtau = Area under the curve from time 0 to 12 hours
Time Frame: Day 4,6,8
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/ml
Groups:
- Dofetilide 500 μg + Placebo (Day 4); Dofetilide 500 μg + Placebo (Day 6); Dofetilide 500 μg +Placebo (Day 8): Dofetilide 500 μg twice a day (BID) orally (Days 1-8) combined to placebo.
- Dofetilide + LQT-1213 (Day 4); Dofetilide + LQT-1213 (Day 6); Dofetilide + LQT-1213 (Day 8): Dofetilide 500 µg twice daily (BID) orally on Days 1-8 and LQT-1213 3 times a day (TID) (0, 7.75, and 17 hours) orally on Days 3-8 as low dose (0.25 mg/kg) on Day 3 through the second dose on Day 4, mid dose (0.50 mg/kg) for last dose on Day 4 through the second dose on Day 6, and high dose (0.70 mg/kg) for last dose on Day 6 through the dose on Day 8.
Arm/Group | Dofetilide 500 μg + Placebo (Day 4) | Dofetilide 500 μg + Placebo (Day 6) | Dofetilide 500 μg +Placebo (Day 8) | Dofetilide + LQT-1213 (Day 4) | Dofetilide + LQT-1213 (Day 6) | Dofetilide + LQT-1213 (Day 8)
Number analyzed (Participants) | 29 | 25 | 25 | 29 | 25 | 25
h*ng/ml | 36.350 (17.3) | 35.916 (15.3) | 37.075 (16.0) | 35.142 (18.4) | 36.390 (16.6) | 38.227 (15.3)

21. Secondary Outcome: Part 1: Pharmacokinetic LQT-1213 Cmax
Description: Maximum observed plasma drug concentration
Time Frame: Day 4,6,8
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: ng/ml
Arm/Group | LQT-1213 0.25 mg/kg (Day 4) TID | LQT-1213 0.50 mg/kg (Day 6) TID | LQT-1213 0.70 mg/kg (Day 8) TID
Number analyzed (Participants) | 29 | 25 | 25
ng/ml | 501.739 (48.0) | 1013.942 (52.1) | 1612.274 (48.5)

22. Secondary Outcome: Part 1: Pharmacokinetic Dofetilide Cmax
Description: Maximum observed plasma drug concentration
Time Frame: Day 4,6, 8
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/ml
Groups:
- Dofetilide 500 μg (Day 4); Dofetilide 500 μg (Day 6); Dofetilide 500 μg (Day 8): Dofetilide 500 μg twice a day (BID) orally (Days 1-8) combined to placebo.
Arm/Group | Dofetilide 500 μg (Day 4) | Dofetilide 500 μg (Day 6) | Dofetilide 500 μg (Day 8) | Dofetilide + LQT-1213 (Day 4) | Dofetilide + LQT-1213 (Day 6) | Dofetilide + LQT-1213 (Day 8)
Number analyzed (Participants) | 29 | 25 | 25 | 29 | 25 | 25
ng/ml | 4.367 (18.7) | 4.394 (16.9) | 4.580 (16.8) | 4.184 (19.0) | 4.438 (19.6) | 4.727 (20.6)

23. Secondary Outcome: Part 1: Pharmacokinetic LQT-1213 Tmax
Description: Time to the maximum observed plasma concentration
Time Frame: Day 4,6,8
Measure: Median (Full Range); unit: hours
Arm/Group | LQT-1213 0.25 mg/kg (Day 4) TID | LQT-1213 0.50 mg/kg (Day 6) TID | LQT-1213 0.70 mg/kg (Day 8) TID
Number analyzed (Participants) | 29 | 25 | 25
hours | 1.012 [0.98 to 6.00] | 1.114 [0.98 to 5.06] | 1.999 [0.99 to 5.05]

24. Secondary Outcome: Part 1: Pharmacokinetic Dofetilide Tmax
Description: Time to the maximum observed plasma concentration
Time Frame: Day 4,6,8
Population: as for outcome 17
Measure: Median (Full Range); unit: hours
Arm/Group | Dofetilide 500 μg (Day 4) | Dofetilide 500 μg (Day 6) | Dofetilide 500 μg (Day 8) | Dofetilide + LQT-1213 (Day 4) | Dofetilide + LQT-1213 (Day 6) | Dofetilide + LQT-1213 (Day 8)
Number analyzed (Participants) | 29 | 25 | 25 | 29 | 25 | 25
hours | 2.012 [1.00 to 6.00] | 2.003 [1.00 to 3.52] | 2.017 [1.00 to 4.01] | 2.015 [1.00 to 451] | 2.008 [1.00 to 5.51] | 2.504 [1.01 to 4.02]

25. Secondary Outcome: Part 1: Pharmacokinetic LQT-1213 t1/2
Description: Terminal half-life
Time Frame: Day 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Groups:
- LQT-1213 TID 0.70 mg/kg: Dofetilide 500 μg BID, orally (Days 1-8) and LQT-1213 TID 0.25 mg/kg (Days 3 and 4), 0.50 mg/kg (Days 5 and 6), and 0.70 mg/kg on (Days 7 and 8). Single dose was given on the morning of Day 8.
Arm/Group | LQT-1213 TID 0.70 mg/kg
Number analyzed (Participants) | 25
hours | 8.374 (22.0)

26. Secondary Outcome: Part 1: Pharmacokinetic Dofetilide t1/2
Description: Terminal half-life
Time Frame: Day 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Dofetilide 500 μg + Placebo Day 8 | Dofetilide + LQT-1213 (Day 8)
Number analyzed (Participants) | 25 | 25
hours | 7.139 (16.2) | 7.341 (14.6)

27. Secondary Outcome: Part 1: Number of Treatment Emerging Adverse Events (TEAEs)
Description: Part 1: Number of Treatment Emerging Adverse Events (TEAEs) that occurred following administration of dofetilide Day1 up to Day 10 period 1 and in period 2 from Day 1 to up to the follow-up visit at Day 17.
Time Frame: Period 1 from Day 1 to Day 10 and Period 2 from Day 1 up to Day 17.
Measure: Number; unit: TEAE
Groups:
- Dofetilide: Dofetilide 500 ug bid Day 1 and Day 2
- Dofetilide + Low Dose LQT-1213 TID 0.25 mg/kg (Days 3 and 4): Dofetilide + LQT-1213 (Low Dose) Day 3 and Day 4
- Dofetilide + Mid Dose LQT-1213 TID 0.50 mg/kg (Days 5 and 6): Dofetilide + LQT-1213 (Mid Dose) Day 5 and Day 6
- Dofetilide + High Dose LQT-1213 TID 0.70 mg/kg (Days 7 and 8): Dofetilide + LQT-1213 (high Dose) Day 7 and Day 8
- Dofetilide + Placebo: Dofetilide + Placebo Day 3 to Day 8
Arm/Group | Dofetilide | Dofetilide + Low Dose LQT-1213 TID 0.25 mg/kg (Days 3 and 4) | Dofetilide + Mid Dose LQT-1213 TID 0.50 mg/kg (Days 5 and 6) | Dofetilide + High Dose LQT-1213 TID 0.70 mg/kg (Days 7 and 8) | Dofetilide + Placebo
Number analyzed (Participants) | 30 | 29 | 29 | 25 | 29
TEAE | 12 | 6 | 12 | 1 | 25

28. Secondary Outcome: Part 2: Pharmacokinetic LQT-1213 AUC0-t
Description: Area under the concentration-time curve (AUC) from time 0 to the time of the last measurable concentration
Time Frame: Day 4 Pre-dose up to 29 hours post-dose administration
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/ml
Arm/Group | LQT-1213 16 mg TID (48 mg Daily) | LQT-1213 7mg Tid (21 mg Daily)
Number analyzed (Participants) | 6 | 6
h*ng/ml | 5968 (30.9) | 2109 (19.5)

29. Secondary Outcome: Part 2: Pharmacokinetic LQT-1213 AUCtau
Description: Pharmacokinetic LQT-1213 AUCtau (time 0 to 8 hours)
Time Frame: day 2 and day 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/ml
Arm/Group | LQT-1213 16 mg TID (48 mg Daily) | LQT-1213 7mg Tid (21 mg Daily)
Number analyzed (Participants) | 6 | 6
h*ng/ml
  Day 2 | 2214 (41.7) | 635.3 (22.8)
  Day 4 | 3314 (32.3) | 1153 (28.0)

30. Secondary Outcome: Part 2: Pharmacokinetic LQT-1213 Cmax
Description: Maximum observed plasma drug concentration
Time Frame: day 2 and day 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/ml
Arm/Group | LQT-1213 16 mg TID (48 mg Daily) | LQT-1213 7mg Tid (21 mg Daily)
Number analyzed (Participants) | 6 | 6
ng/ml
  Day 2 | 470.9 (46.5) | 116.4 (23.8)
  Day 4 | 562.9 (44.4) | 195.1 (33.9)

31. Secondary Outcome: Part 2: Pharmacokinetic LQT-1213 Tmax
Description: Time to the maximum observed plasma concentration
Time Frame: Day 2 and Day 4
Measure: Median (Full Range); unit: ng/ml
Arm/Group | LQT-1213 16 mg TID (48 mg Daily) | LQT-1213 7mg Tid (21 mg Daily)
Number analyzed (Participants) | 6 | 6
ng/ml
  Day 2 | 1.523 [1.01 to 4.01] | 1.268 [1.00 to 2.01]
  Day 4 | 1.534 [0.98 to 4.01] | 1.781 [1.02 to 5.00]

32. Secondary Outcome: Part 2: Pharmacokinetic LQT-1213 t1/2
Description: Part 2: Pharmacokinetic LQT-1213 terminal half-life t1/2
Time Frame: Day 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | LQT-1213 16 mg TID (48 mg Daily) | LQT-1213 7mg Tid (21 mg Daily)
Number analyzed (Participants) | 6 | 6
hours | 11.97 (11.8) | 9.982 (9.8)

33. Other Pre Specified Outcome: Part 2: Time-matched Placebo-corrected QTcF - 1 Hour Post Dose
Description: QTcF values at each timepoint on Days 4 were compared to the time-matched QTcF values on Day 1 (placebo) using the paired t-test.
Time Frame: 1 hour after administration of study treatment on Day 4.
Measure: Mean (Standard Deviation); unit: msec
Groups:
- LQT-1213 16 mg TID (48 mg Daily) Day 4: LQT-1213 16 mg TID (at time 0, 8 and 16 hours) on Days 2-4, with a final single morning dose on Day 4.
- Placebo TID (Day1): Day 1 was placebo TID.
Arm/Group | LQT-1213 16 mg TID (48 mg Daily) Day 4 | Placebo TID (Day1)
Number analyzed (Participants) | 6 | 6
msec | 519.17 (32.344) | 514.89 (29.569)
Statistical Analysis 1: Comparison: LQT-1213 16 mg TID (48 mg Daily) Day 4 vs Placebo TID (Day1); Test type: Superiority; p = 0.3169, t-test, 2 sided; Mean Difference (Net) = 4.28

34. Other Pre Specified Outcome: Part 2: Time-matched Placebo-corrected QTcF at 2 Hours Post-dose
Description: QTcF values at each timepoint on Day 4 were compared to the time-matched QTcF value on Day 1 (placebo) using the paired t-test.
Time Frame: 2 hours after administration of study treatment on Day 4.
Measure: Mean (Standard Deviation); unit: msec
Groups:
- TID Dosing of LQT-1213 16 mg Day 4 (48 mg Daily): LQT-1213 16 mg TID (at time 0, 8 and 16 hours) on Days 2-4, with a final single morning dose on Day 4.
- TID Dosing of Placebo (Day 1): TID dosing of placebo (Day 1).
Arm/Group | TID Dosing of LQT-1213 16 mg Day 4 (48 mg Daily) | TID Dosing of Placebo (Day 1)
Number analyzed (Participants) | 6 | 6
msec | 520.06 (31.231) | 513.28 (23.733)
Statistical Analysis 1: Comparison: TID Dosing of LQT-1213 16 mg Day 4 (48 mg Daily) vs TID Dosing of Placebo (Day 1); Test type: Superiority; p = 0.1066, t-test, 2 sided; Mean Difference (Net) = 6.78

35. Other Pre Specified Outcome: Part 2: Time-matched Placebo-corrected QTcF at 3 Hours Post-dose
Description: as for outcome 33
Time Frame: 3 hours after administration of study treatment on Day 4.
Measure: Mean (Standard Deviation); unit: msec
Groups:
- Placebo TID Dosing Day 1: Placebo TID Dosing Day 1.
Arm/Group | TID Dosing of LQT-1213 16 mg Day 4 (48 mg Daily) | Placebo TID Dosing Day 1
Number analyzed (Participants) | 6 | 6
msec | 513.94 (26.410) | 530.00 (39.838)
Statistical Analysis 1: Comparison: TID Dosing of LQT-1213 16 mg Day 4 (48 mg Daily) vs Placebo TID Dosing Day 1; Test type: Superiority; p = 0.0443, t-test, 2 sided; Mean Difference (Net) = -16.06

36. Other Pre Specified Outcome: Part 2: Time-matched Placebo-corrected QTcF at 4 Hours Post-dose
Description: as for outcome 33
Time Frame: 4 hours after administration of study treatment on Day 4.
Measure: Mean (Standard Deviation); unit: msec
Groups:
- TID Dosing of LQT-1213 16 mg Day 4 (48 mg Daily): LQT-1213 16 mg TID (at time 0, 8 and 16 hours) on Days 2-4, with a final single morning dose on Day 4. Day 1 was placebo.
Arm/Group | TID Dosing of LQT-1213 16 mg Day 4 (48 mg Daily) | TID Dosing of Placebo (Day 1)
Number analyzed (Participants) | 6 | 6
msec | 514.61 (28.450) | 523.67 (32.158)
Statistical Analysis 1: Comparison: TID Dosing of LQT-1213 16 mg Day 4 (48 mg Daily) vs TID Dosing of Placebo (Day 1); Test type: Superiority; p = 0.0815, t-test, 2 sided; Mean Difference (Net) = -9.06

37. Other Pre Specified Outcome: Part 2: Time-matched Placebo-corrected QTcF at 6 Hours Post-dose
Description: as for outcome 33
Time Frame: 6 hours after administration of study treatment on Day 4.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | TID Dosing of LQT-1213 16 mg Day 4 (48 mg Daily) | TID Dosing of Placebo (Day 1)
Number analyzed (Participants) | 6 | 6
msec | 520.89 (26.741) | 531.56 (32.897)
Statistical Analysis 1: Comparison: TID Dosing of LQT-1213 16 mg Day 4 (48 mg Daily) vs TID Dosing of Placebo (Day 1); Test type: Superiority; p = 0.0137, t-test, 2 sided; Mean Difference (Net) = -10.67

38. Other Pre Specified Outcome: Part 2: Time-matched Placebo-corrected QTcF at 8 Hours Post-dose
Description: as for outcome 33
Time Frame: 8 hours after administration of study treatment on Day 4.
Measure: Mean (Standard Deviation); unit: msec
Groups:
- TID Dosing Placebo (Day 1): TID Dosing Placebo (Day 1)
Arm/Group | TID Dosing of LQT-1213 16 mg Day 4 (48 mg Daily) | TID Dosing Placebo (Day 1)
Number analyzed (Participants) | 6 | 6
msec | 503.61 (22.106) | 507.61 (23.640)
Statistical Analysis 1: Comparison: TID Dosing of LQT-1213 16 mg Day 4 (48 mg Daily) vs TID Dosing Placebo (Day 1); Test type: Superiority; p = 0.3539, t-test, 2 sided; Mean Difference (Net) = -4.00

39. Other Pre Specified Outcome: Part 2: Time-matched Placebo-corrected QTcF at 10 Hours Post-dose
Description: as for outcome 33
Time Frame: 10 hours after administration of study treatment on Day 4.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | TID Dosing of LQT-1213 16 mg Day 4 (48 mg Daily) | TID Dosing Placebo (Day 1)
Number analyzed (Participants) | 6 | 6
msec | 521.00 (9.78) | 511.22 (22.872)
Statistical Analysis 1: Comparison: TID Dosing of LQT-1213 16 mg Day 4 (48 mg Daily) vs TID Dosing Placebo (Day 1); Test type: Superiority; p = 0.1377, t-test, 2 sided; Mean Difference (Net) = 9.78

40. Other Pre Specified Outcome: Part 2: Time-matched Placebo-corrected QTcF at 12 Hours Post-dose
Description: as for outcome 33
Time Frame: 12 hours after administration of study treatment on Day 4.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | TID Dosing of LQT-1213 16 mg Day 4 (48 mg Daily) | TID Dosing Placebo (Day 1)
Number analyzed (Participants) | 6 | 6
msec | 519.42 (26.753) | 522.11 (23.167)
Statistical Analysis 1: Comparison: TID Dosing of LQT-1213 16 mg Day 4 (48 mg Daily) vs TID Dosing Placebo (Day 1); Test type: Superiority; p = 0.6184, t-test, 2 sided; Mean Difference (Net) = -2.69

41. Other Pre Specified Outcome: Part 2: Time-matched Placebo-corrected QTcF at 1 Hour Post-dose (Low Dose)
Description: as for outcome 33
Time Frame: 1 hours after administration of study treatment on Day 4.
Measure: Mean (Standard Deviation); unit: msec
Groups:
- TID Dosing of LQT-1213 7 mg Day 4 (21 mg Daily): LQT-1213 7 mg TID (at time 0, 8 and 16 hours) on Days 2-4, with a final single morning dose on Day 4.
- TID Dosing Placebo Day 1: TID Dosing Placebo Day 1.
Arm/Group | TID Dosing of LQT-1213 7 mg Day 4 (21 mg Daily) | TID Dosing Placebo Day 1
Number analyzed (Participants) | 6 | 6
msec | 524.39 (29.611) | 521.22 (33.791)
Statistical Analysis 1: Comparison: TID Dosing of LQT-1213 7 mg Day 4 (21 mg Daily) vs TID Dosing Placebo Day 1; Test type: Superiority; p = 0.6627, t-test, 2 sided; Mean Difference (Net) = 3.17

42. Other Pre Specified Outcome: Part 2: Time-matched Placebo-corrected QTcF at 2 Hours Post-dose (Low Dose)
Description: as for outcome 33
Time Frame: 2 hours after administration of study treatment on Day 4.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | TID Dosing of LQT-1213 7 mg Day 4 (21 mg Daily) | TID Dosing Placebo Day 1
Number analyzed (Participants) | 6 | 6
msec | 531.72 (38.880) | 525.94 (29.837)
Statistical Analysis 1: Comparison: TID Dosing of LQT-1213 7 mg Day 4 (21 mg Daily) vs TID Dosing Placebo Day 1; Test type: Superiority; p = 0.5276, t-test, 2 sided; Mean Difference (Net) = 5.78

43. Other Pre Specified Outcome: Part 2: Time-matched Placebo-corrected QTcF at 3 Hours Post-dose (Low Dose)
Description: QTcF values at each timepoint on Days 4 were compared to the time-matched QTcF values on Day 1 (placebo) using the paired t-test, which was the same as analyzing the difference of the time-matched QTcF values using one-sample t test.
Time Frame: 3 hours after administration of study treatment on Day 4.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | TID Dosing of LQT-1213 7 mg Day 4 (21 mg Daily) | TID Dosing Placebo Day 1
Number analyzed (Participants) | 6 | 6
msec | 538.22 (38.584) | 523.06 (33.857)
Statistical Analysis 1: Comparison: TID Dosing of LQT-1213 7 mg Day 4 (21 mg Daily) vs TID Dosing Placebo Day 1; Test type: Superiority; p = 0.0399, t-test, 2 sided; Mean Difference (Net) = 15.17

44. Other Pre Specified Outcome: Part 2: Time-matched Placebo-corrected QTcF at 4 Hours Post-dose (Low Dose)
Description: as for outcome 33
Time Frame: 4 hours after administration of study treatment on Day 4.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | TID Dosing of LQT-1213 7 mg Day 4 (21 mg Daily) | TID Dosing Placebo Day 1
Number analyzed (Participants) | 6 | 6
msec | 535.72 (34.812) | 522.17 (35.036)
Statistical Analysis 1: Comparison: TID Dosing of LQT-1213 7 mg Day 4 (21 mg Daily) vs TID Dosing Placebo Day 1; Test type: Superiority; p = 0.0747, t-test, 2 sided; Mean Difference (Net) = 13.56

45. Other Pre Specified Outcome: Part 2: Time-matched Placebo-corrected QTcF at 6 Hours Post-dose (Low Dose)
Description: as for outcome 33
Time Frame: 6 hours after administration of study treatment on Day 4.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | TID Dosing of LQT-1213 7 mg Day 4 (21 mg Daily) | TID Dosing Placebo Day 1
Number analyzed (Participants) | 6 | 6
msec | 530.67 (43.213) | 530.17 (32.590)
Statistical Analysis 1: Comparison: TID Dosing of LQT-1213 7 mg Day 4 (21 mg Daily); Test type: Superiority; p = 0.9584, t-test, 2 sided

46. Other Pre Specified Outcome: Part 2: Time-matched Placebo-corrected QTcF at 8 Hours Post-dose (Low Dose)
Description: as for outcome 33
Time Frame: 8 hours after administration of study treatment on Day 4.
Measure: Mean (Standard Deviation); unit: msec
Groups:
- TID Dosing of LQT-1213 7 mg (21 mg Daily): LQT-1213 7 mg TID (at time 0, 8 and 16 hours) on Days 2-4, with a final single morning dose on Day 4. Day 1 was placebo.
Arm/Group | TID Dosing of LQT-1213 7 mg (21 mg Daily) | TID Dosing Placebo Day 1
Number analyzed (Participants) | 6 | 6
msec | 522.67 (33.363) | 516.94 (51.848)
Statistical Analysis 1: Comparison: TID Dosing of LQT-1213 7 mg (21 mg Daily) vs TID Dosing Placebo Day 1; Test type: Superiority; p = 0.6531, t-test, 2 sided; Mean Difference (Net) = 5.72

47. Other Pre Specified Outcome: Part 2: Time-matched Placebo-corrected QTcF at 10 Hours Post-dose (Low Dose)
Description: as for outcome 33
Time Frame: 10 hours after administration of study treatment on Day 4.
Measure: Mean (Standard Deviation); unit: msec
Groups:
- TID Dosing of LQT-1213 7 mg Day 4 (21 mg Daily): LQT-1213 7 mg TID (at time 0, 8 and 16 hours) on Days 2-4, with a final single morning dose on Day 4. Day 1 was placebo.
Arm/Group | TID Dosing of LQT-1213 7 mg Day 4 (21 mg Daily) | TID Dosing Placebo Day 1
Number analyzed (Participants) | 6 | 6
msec | 530.39 (40.667) | 514.78 (38.749)
Statistical Analysis 1: Comparison: TID Dosing of LQT-1213 7 mg Day 4 (21 mg Daily) vs TID Dosing Placebo Day 1; Test type: Superiority; p = 0.0482, t-test, 2 sided; Mean Difference (Net) = 15.61

48. Other Pre Specified Outcome: Part 2: Time-matched Placebo-corrected QTcF at 12 Hours Post-dose (Low Dose)
Description: as for outcome 33
Time Frame: 12 hours after administration of study treatment on Day 4.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | TID Dosing of LQT-1213 7 mg Day 4 (21 mg Daily) | TID Dosing Placebo Day 1
Number analyzed (Participants) | 6 | 6
msec | 536.11 (44.465) | 518.89 (39.724)
Statistical Analysis 1: Comparison: TID Dosing of LQT-1213 7 mg Day 4 (21 mg Daily) vs TID Dosing Placebo Day 1; Test type: Superiority; p = 0.0667, t-test, 2 sided; Mean Difference (Net) = 17.22

49. Other Pre Specified Outcome: Part 2: ΔAUC2-6 Hours QTcF Values on Day 4 (LQT-1213 16 mg TID) Compared to the Time-matched on Day 1 (Placebo)
Description: QTcF area under the curve on Day 4 (2 to 6 hours; LQT-1213) was compared to QTcF AUC on Day 1 (2 to 6 hours; placebo).
Time Frame: Day 4
Measure: Mean (Standard Deviation); unit: msec*hour
Groups:
- TID Dosing of Placebo Day1: TID Dosing of Placebo Day1.
Arm/Group | TID Dosing of Placebo Day1 | TID Dosing of LQT-1213 16 mg Day 4 (48 mg Daily)
Number analyzed (Participants) | 6 | 6
msec*hour | 2103.69 (130.872) | 2066.69 (113.850)
Statistical Analysis 1: Comparison: TID Dosing of Placebo Day1 vs TID Dosing of LQT-1213 16 mg Day 4 (48 mg Daily); Test type: Superiority; p = 0.0131, t-test, 2 sided; Mean Difference (Net) = -37.00

50. Other Pre Specified Outcome: Part 2: ΔAUC3-6 Hours QTcF Values on Day 4 (LQT-1213 16 mg TID) Compared to the Time-matched on Day 1 (Placebo)
Description: QTcF area under the curve on Day 4 (3 to 6 hours; LQT-1213) was compared to QTcF AUC on Day 1 (3 to 6 hours; placebo).
Time Frame: Day 4
Measure: Mean (Standard Deviation); unit: msec*hour
Arm/Group | TID Dosing of Placebo Day1 | TID Dosing of LQT-1213 16 mg Day 4 (48 mg Daily)
Number analyzed (Participants) | 6 | 6
msec*hour | 1582.06 (100.213) | 1549.69 (85.553)
Statistical Analysis 1: Comparison: TID Dosing of Placebo Day1 vs TID Dosing of LQT-1213 16 mg Day 4 (48 mg Daily); Test type: Superiority; p = 0.0141, t-test, 2 sided; Mean Difference (Net) = -32.36

51. Other Pre Specified Outcome: Part 2: ΔAUC0-8 Hours QTcF Values on Day 4 (LQT-1213 16 mg TID) Compared to the Time-matched on Day 1 (Placebo)
Description: QTcF area under the curve on Day 4 (0 to 8 hours; LQT-1213) was compared to QTcF AUC on Day 1 (0 to 8 hours; placebo).
Time Frame: Day 4
Measure: Mean (Standard Deviation); unit: msec*hour
Arm/Group | TID Dosing of Placebo Day1 | TID Dosing of LQT-1213 16 mg Day 4 (48 mg Daily)
Number analyzed (Participants) | 6 | 6
msec*hour | 4173.19 (236.787) | 4128.64 (224.746)
Statistical Analysis 1: Comparison: TID Dosing of Placebo Day1 vs TID Dosing of LQT-1213 16 mg Day 4 (48 mg Daily); Test type: Superiority; p = 0.0019, t-test, 2 sided; Mean Difference (Net) = -44.55

52. Other Pre Specified Outcome: Part 2: ΔAUC0-12 Hours QTcF Values on Day 4 (LQT-1213 16 mg TID) Compared to the Time-matched on Day 1 (Placebo)
Description: QTcF area under the curve on Day 4 (0 to 12 hours; LQT-1213) was compared to QTcF AUC on Day 1 (0 to 12 hours; placebo).
Time Frame: Day 4
Measure: Mean (Standard Deviation); unit: msec*hour
Arm/Group | TID Dosing of Placebo Day1 | TID Dosing of LQT-1213 16 mg Day 4 (48 mg Daily)
Number analyzed (Participants) | 6 | 6
msec*hour | 6225.35 (323.651) | 6193.67 (314.325)
Statistical Analysis 1: Comparison: TID Dosing of Placebo Day1 vs TID Dosing of LQT-1213 16 mg Day 4 (48 mg Daily); Test type: Superiority; p = 0.1108, t-test, 2 sided; Mean Difference (Net) = -31.69

53. Other Pre Specified Outcome: Part 2: ΔAUC2-6 Hours QTcF Values on Day 4 (LQT-1213 7 mg TID) Compared to the Time-matched on Day 1 (Placebo)
Description: QTcF area under the curve on Day 4 (2 to 6 hours; LQT-1213) was compared to QTcF AUC on Day 1 (2 to 6 hours; placebo).
Time Frame: Day 4
Measure: Mean (Standard Deviation); unit: msec*hour
Arm/Group | TID Dosing of Placebo Day1 | TID Dosing of LQT-1213 7 mg Day 4 (21 mg Daily)
Number analyzed (Participants) | 6 | 6
msec*hour | 2099.44 (132.566) | 2137.25 (150.766)
Statistical Analysis 1: Comparison: TID Dosing of Placebo Day1 vs TID Dosing of LQT-1213 7 mg Day 4 (21 mg Daily); Test type: Superiority; p = 0.1840, t-test, 2 sided; Mean Difference (Net) = 37.81

54. Other Pre Specified Outcome: Part 2: ΔAUC3-6 Hours QTcF Values on Day 4 (LQT-1213 7 mg TID) Compared to the Time-matched on Day 1 (Placebo)
Description: QTcF area under the curve on Day 4 (3 to 6 hours; LQT-1213) was compared to QTcF AUC on Day 1 (3 to 6 hours; placebo).
Time Frame: Day 4
Measure: Mean (Standard Deviation); unit: msec*hour
Arm/Group | TID Dosing of Placebo Day1 | TID Dosing of LQT-1213 7 mg (21 mg Daily)
Number analyzed (Participants) | 6 | 6
msec*hour | 1574.94 (101.583) | 1602.28 (112.284)
Statistical Analysis 1: Comparison: TID Dosing of Placebo Day1 vs TID Dosing of LQT-1213 7 mg (21 mg Daily); Test type: Superiority; p = 0.2019, t-test, 2 sided; Mean Difference (Net) = 27.33

55. Other Pre Specified Outcome: Part 2: ΔAUC0-8 Hours QTcF Values on Day 4 (LQT-1213 7 mg TID) Compared to the Time-matched on Day 1 (Placebo)
Description: QTcF area under the curve on Day 4 (0 to 8 hours; LQT-1213) was compared to QTcF AUC on Day 1 (0 to 8 hours; placebo).
Time Frame: Day 4
Measure: Mean (Standard Deviation); unit: msec*hour
Arm/Group | TID Dosing of Placebo Day1 | TID Dosing of LQT-1213 7 mg Day 4 (21 mg Daily)
Number analyzed (Participants) | 6 | 6
msec*hour | 4192.47 (279.304) | 4248.69 (290.144)
Statistical Analysis 1: Comparison: TID Dosing of LQT-1213 7 mg Day 4 (21 mg Daily); Test type: Superiority; p = 0.2808, t-test, 2 sided

56. Other Pre Specified Outcome: Part 2: ΔAUC0-12 Hours QTcF Values on Day 4 (LQT-1213 7 mg TID) Compared to the Time-matched on Day 1 (Placebo)
Description: QTcF area under the curve on Day 4 (0 to 12 hours; LQT-1213) was compared to QTcF AUC on Day 1 (0 to 12 hours; placebo).
Time Frame: Day 4
Measure: Mean (Standard Deviation); unit: msec*hour
Arm/Group | TID Dosing of Placebo Day1 | TID Dosing of LQT-1213 7 mg (21 mg Daily)
Number analyzed (Participants) | 6 | 6
msec*hour | 6257.86 (445.699) | 6368.25 (444.031)
Statistical Analysis 1: Comparison: TID Dosing of Placebo Day1 vs TID Dosing of LQT-1213 7 mg (21 mg Daily); Test type: Superiority; p = 0.1644, t-test, 2 sided; Mean Difference (Net) = 110.39

57. Other Pre Specified Outcome: Part 2: ΔAUC2-6 Hours QTcF Values on Day 4 (LQT-1213 16 mg TID) Compared to the Time-matched on Day 1 (Placebo) Subgroup Analysis (≥ 500ms)
Description: QTcF area under the curve on Day 4 (2 to 6 hours; LQT-1213) was compared to QTcF AUC on Day 1 (2 to 6 hours; placebo) for subjects with a Day 1 Pre-Dose (Baseline 1) QTcF >= 500 ms
Time Frame: Day 4
Measure: Mean (Standard Deviation); unit: msec*hour
Arm/Group | TID Dosing of Placebo Day1 | TID Dosing of LQT-1213 16 mg Day 4 (48 mg Daily)
Number analyzed (Participants) | 4 | 4
msec*hour | 2175.83 (85.532) | 2131.54 (69.025)
Statistical Analysis 1: Comparison: TID Dosing of Placebo Day1 vs TID Dosing of LQT-1213 16 mg Day 4 (48 mg Daily); Test type: Superiority; p = 0.0282, t-test, 2 sided; Mean Difference (Net) = -44.29

58. Other Pre Specified Outcome: Part 2: ΔAUC3-6 Hours QTcF Values on Day 4 (LQT-1213 16 mg TID) Compared to the Time-matched on Day 1 (Placebo) Subgroup Analysis (≥ 500ms)
Description: QTcF area under the curve on Day 4 (3 to 6 hours; LQT-1213) was compared to QTcF AUC on Day 1 (3 to 6 hours; placebo) for subjects with a Day 1 Pre-Dose (Baseline 1) QTcF >= 500 ms
Time Frame: Day 4
Measure: Mean (Standard Deviation); unit: msec*hour
Arm/Group | TID Dosing of Placebo Day1 | TID Dosing of LQT-1213 16 mg Day 4 (48 mg Daily)
Number analyzed (Participants) | 4 | 4
msec*hour | 1636.33 (68.013) | 1598.46 (51.804)
Statistical Analysis 1: Comparison: TID Dosing of Placebo Day1 vs TID Dosing of LQT-1213 16 mg Day 4 (48 mg Daily); Test type: Superiority; p = 0.0306, t-test, 2 sided; Mean Difference (Net) = -37.87

59. Other Pre Specified Outcome: Part 2: ΔAUC0-8 Hours QTcF Values on Day 4 (LQT-1213 16 mg TID) Compared to the Time-matched on Day 1 (Placebo) Subgroup Analysis (≥ 500ms)
Description: QTcF area under the curve on Day 4 (0 to 8 hours; LQT-1213) was compared to QTcF AUC on Day 1 (0 to 8 hours; placebo) for subjects with a Day 1 Pre-Dose (Baseline 1) QTcF >= 500 ms
Time Frame: Day 4
Measure: Mean (Standard Deviation); unit: msec*hour
Arm/Group | TID Dosing of Placebo Day1 | TID Dosing of LQT-1213 16 mg Day 4 (48 mg Daily)
Number analyzed (Participants) | 4 | 4
msec*hour | 4308.79 (135.627) | 4255.38 (138.707)
Statistical Analysis 1: Comparison: TID Dosing of Placebo Day1 vs TID Dosing of LQT-1213 16 mg Day 4 (48 mg Daily); Test type: Superiority; p = 0.0016, t-test, 2 sided; Mean Difference (Net) = -53.42

60. Other Pre Specified Outcome: Part 2: ΔAUC0-12 Hours QTcF Values on Day 4 (LQT-1213 16 mg TID) Compared to the Time-matched on Day 1 (Placebo) Subgroup Analysis (≥ 500ms)
Description: QTcF area under the curve on Day 4 (0 to 12 hours; LQT-1213) was compared to QTcF AUC on Day 1 (0 to 12 hours; placebo) for subjects with a Day 1 Pre-Dose (Baseline 1) QTcF >= 500 ms
Time Frame: Day 4
Measure: Mean (Standard Deviation); unit: msec*hour
Arm/Group | TID Dosing of Placebo Day1 | TID Dosing of LQT-1213 16 mg Day 4 (48 mg Daily)
Number analyzed (Participants) | 4 | 4
msec*hour | 6413.29 (175.189) | 6369.04 (200.818)
Statistical Analysis 1: Comparison: TID Dosing of LQT-1213 16 mg Day 4 (48 mg Daily); Test type: Superiority; p = 0.1378, t-test, 2 sided; Mean Difference (Net) = -44.25

ADVERSE EVENTS:
Time Frame: Part 1 : Period 1 (Day 1 to Day 10) and Period 2 (Day 1 to Day 17). Part 2: 12 days
Groups:
- Dofetilide + Low Dose LQT-1213 TID 0.25 mg/kg (Days 3 and 4): Dofetilide + Low dose LQT-1213 TID 0.25 mg/kg (Days 3 and 4)
- Dofetilide + Mid Dose LQT-1213 TID 0.50 mg/kg (Days 5 and 6): Dofetilide + Mid dose LQT-1213 TID 0.50 mg/kg (Days 5 and 6)
- Dofetilide + High Dose LQT-1213 0.70 mg/kg on (Days 7 and 8): Dofetilide + High Dose LQT-1213 0.70 mg/kg on (Days 7 and 8)
- LQT-1213 16 mg TID: LQT-1213 16 mg TID Day 2 to Day 4 (48 mg Daily)
- LQT-1213 7 mg TID: LQT-1213 7 mg TID Day 2 to Day 4 (21 mg Daily)
- Placebo Matching LQT-1213 16 mg TID: Placebo matching LQT-1213 16 mg TID (Day 1)
- Placebo Matching LQT-1213 7 mg TID: Placebo matching LQT-1213 7 mg TID (Day 1)
Arm/Group | Dofetilide | Dofetilide + Low Dose LQT-1213 TID 0.25 mg/kg (Days 3 and 4) | Dofetilide + Mid Dose LQT-1213 TID 0.50 mg/kg (Days 5 and 6) | Dofetilide + High Dose LQT-1213 0.70 mg/kg on (Days 7 and 8) | Dofetilide + Placebo | LQT-1213 16 mg TID | LQT-1213 7 mg TID | Placebo Matching LQT-1213 16 mg TID | Placebo Matching LQT-1213 7 mg TID
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/29 | 0/29 | 0/25 | 0/25 | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/29 | 0/29 | 0/25 | 0/29 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/30 | 0/29 | 2/29 | 0/25 | 4/29 | 3/6 | 1/6 | 1/6 | 2/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dofetilide (N=30) | Dofetilide + Low Dose LQT-1213 TID 0.25 mg/kg (Days 3 and 4) (N=29) | Dofetilide + Mid Dose LQT-1213 TID 0.50 mg/kg (Days 5 and 6) (N=29) | Dofetilide + High Dose LQT-1213 0.70 mg/kg on (Days 7 and 8) (N=25) | Dofetilide + Placebo (N=29) | LQT-1213 16 mg TID (N=6) | LQT-1213 7 mg TID (N=6) | Placebo Matching LQT-1213 16 mg TID (N=6) | Placebo Matching LQT-1213 7 mg TID (N=6)
Vessel puncture site pain (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Skin tightness (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Skin warm (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinitis atrophic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Electrode site irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-12-05): https://cdn.clinicaltrials.gov/large-docs/32/NCT05906732/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-19): https://cdn.clinicaltrials.gov/large-docs/32/NCT05906732/SAP_001.pdf